CLINICAL TRIAL: NCT03382028
Title: Development of Child With Equinus Deformity Idiopathic
Acronym: DENEBO1
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_3061-DENEBO1; 2016-A01975-46 (Other: committee for the protection of persons ile de france III)
Record Dates: First submitted 2017-11-16; First posted 2017-12-22 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-11

CONDITIONS: Equinus Deformity
Keywords: developmental abnormalities; psychomotor development
MeSH Terms: conditions — Equinus Deformity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Identification and characterization of the link between psychomotor development and the appearance of associated signs in children with "Equinus Deformity " considered isolated at birth.

DETAILED DESCRIPTION:
The main objective of this study is to define the frequency of developmental abnormalities in children with "Equinus Deformity Idiopathic" compared to the general population

The secondary objective is to identify the prenatal and / or neonatal characteristics that could be predictive of the occurrence of developmental abnormalities in

Prenatal and postnatal follow-up data are derived from the child's medical file. To complete these data and after inclusion, parents of children carrying "Equinus Deformity Idiopathic" will be sent a questionnaire that assesses overall psychomotor development and lists the medical events since the birth of their child (scoliosis, epilepsy ...).

ELIGIBILITY:
Inclusion Criteria:

* Children born between January 2002 and August 2015
* Prenatal or postnatal diagnosis of idiopathic or syndromic Equinus Deformity
* Followed by the pediatric orthopedic service of Rennes University Hospital
* Parent having received the information on the protocol and having not expressed their opposition.

Exclusion Criteria:

* Parents opposing the study

Ages: 2 Years to 15 Years | Sex: All
Age Groups: Child
Gender Based: Yes
Study Population: Children with Equinus Deformity
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Frequency of developmental abnormalities (with the exception of Equinus Deformity) in children with Equinus Deformity idiopathic compared to the general population. | through study completion an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Pasquier, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, France

IPD SHARING:
Plan to Share IPD: No